CLINICAL TRIAL: NCT02114957
Title: Single Oral Dose Pharmacokinetics of Decursin/Decursinol Angelate in Healthy Adult Men and Women
Brief Title: Pharmacokinetics of Decursin/Decursinol Angelate (CognIQTM)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A12-3742
Record Dates: First submitted 2014-04-11; First posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
Keywords: bio-availability; decursin; decursinol angelate; decursinol; subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- study herb (Experimental)
  Interventions: Dietary Supplement: 800mg dietary supplement CognIQTM (4 capsules) by oral at hour 0

INTERVENTIONS:
Dietary Supplement: 800mg dietary supplement CognIQTM (4 capsules) by oral at hour 0

SUMMARY:
This study is to investigate how human bodies absorb and metabolize two herbal drugs. The information is critical for drug development and could not be obtained from any other studies using animals. The two herbal drugs are decursin and decursinol angelate (DA) which naturally exist in a traditional herb Angelica gigas Nakai (AGN). Preclinical and clinical studies indicated that AGN and decursin/DA were quite safe to animals and human.

ELIGIBILITY:
Inclusion Criteria:

* Health subjects weighing between 50 to 91 kilograms (110 to 200 pounds)
* Subjects 18 to 65 years of age
* Subjects having normal hepatic, renal and bone marrow function as assessed by history, physical and clinical chemistry analysis

Exclusion Criteria:

* Subjects positive for HIV, HBV and HCV
* Subjects with diabetes-due to length of fasting
* Subjects regularly taking any kind of prescription medications
* Subjects taking oral contraception, hormone-containing IUDs, contraception implants, or Depo medroxyprogesterone injections
* Subjects taking any food or herbal supplements containing AGN (e.g. CognIQTM, D-Cursinol, Decursinol-50™, Ache Action™, Fast-Acting Joint Formula, EstroG-100™) within 30 days of the study.
* Female subjects that are pregnant, <6 months postpartum, or breastfeeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of decursin, decursinol angelate (DA) and decursinol | 0, 0.5, 1, 2, 3, 4, 6, 8, 12 , 24, 48 hours post-dose

SECONDARY OUTCOMES:
vital signs, plasma biochemistry and blood cell counts of subjects after consumption the study herb | 0 and 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Jinhui Zhang, Ph.D, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Clinical Research Unit, School of Medicine, Texas Tech University Health Sciences Center, Amarillo, Texas, United States

REFERENCES:
- [Derived] Zhang J, Li L, Hale TW, Chee W, Xing C, Jiang C, Lu J. Single oral dose pharmacokinetics of decursin and decursinol angelate in healthy adult men and women. PLoS One. 2015 Feb 19;10(2):e0114992. doi: 10.1371/journal.pone.0114992. eCollection 2015. PMID 25695490